CLINICAL TRIAL: NCT05487326
Title: Comparison of Pain Relief Between High Thoracic Erector Spinae Plane Block and Cervical Epidural Injection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, Ji Hee Hong, Professor, Keimyung University Dongsan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-01-026-03
Record Dates: First submitted 2022-08-01; First posted 2022-08-04 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Pain, Chronic
Keywords: Pain, lumbar
MeSH Terms: conditions — Chronic Pain; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high thoracic ESPB group (Active Comparator): Group where ESPB is performed at T2 with local anesthetic mixture 20 ml
  Interventions: Procedure: Erector spinae plane block
- cervical epidural group (Active Comparator): Group where cervical epidural injection is performed at C6-7 or C7-T1 level
  Interventions: Procedure: cervical epidural injection

INTERVENTIONS:
Procedure: Erector spinae plane block — fascial plane injection guided by ultrasound guidance
  Arms: high thoracic ESPB group
Procedure: cervical epidural injection — cervical epidural injection by fluoroscopy
  Arms: cervical epidural group

SUMMARY:
The primary endpoint of this study was to identify whether there is a pain improving effect of high thoracic eretor spinae plane block (ESPB) when compared with cervical epidural injection

DETAILED DESCRIPTION:
The erector spinae plane block (ESPB) is a less invasive, safer, and technically easy alternative procedure to conventional neuraxial anesthetic techniques. In contrast to common neuraxial techniques such as paravertebral and epidural injections, the ESPB targets an interfascial plane which is far from the spinal cord, root, and pleura. First applied to thoracic neuropathic pain, currently ESPB is being applied to postoperative pain control and includes variable clinical situations. In the abdomen and thoracic wall, thoracic ESPB can be applied for pain control after cardiac surgery, video-assisted thoracic surgery, laparoscopic cholecystectomy, and thoracotomy. Recently, favorable postoperative pain control after lumbar spinal or lower limb surgeries has been reported with lumbar ESPB. In addition, ESPB has also been used for chronic pain conditions in the upper and lower extremities. To investigate the possible mechanism of action of the ESPB, many previous studies have focused on examining the physical spread of the injected agent. Commonly, contrast dye injections in human cadavers have been utilized to assess the spread level. Physical spread level was determined using various methods including direct dissection or sectioning, computed tomography (CT), thoracoscopic inspection, or magnetic resonance imaging (MRI) with radiocontrast injection. Apart from human cadaver studies, physical spread level has been evaluated in alive patients using a variable volume of local anesthetics mixed with radiocontrast. However, these studies are limited by the small number of included patients.

ELIGIBILITY:
Inclusion Criteria:

* cervical spinal stenosis
* cervical intervertebral disc herniation
* cervical facet arthropathy
* cervical foraminal stenosis

Exclusion Criteria:

* Allergy to local anesthetics or contrast medium
* Pregnancy
* Spine deformity
* Patients with coagulation abnormality

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2022-08-07 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Changes of numerical rating scale | baseline, 10 min after injection, 1wk after injection, 2 wks after injection, 4 wks after injection, 8 wks after injection
  Changes of 11-point numerical rating scale (0-10)

SECONDARY OUTCOMES:
Changes of neck disability index | baseline, 8 wks after injection
  Changes of back pain funtional scale

CONTACTS AND LOCATIONS:
Overall Officials: Ji H Hong, Ph.D, Principal Investigator — Keimyung University
Locations (1):
- Hong ji HEE, Daegu, South Korea